CLINICAL TRIAL: NCT00481533
Title: Prophylactic Ergonovine-Oxytocin Versus Oxytocin During Cesarean Delivery Following Failure to Progress in Labour
Brief Title: Ergot and Oxytocin During Cesarean Delivery Following Failure to Progress in Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-07; 05-0042-A
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Blood Loss, Surgical
Keywords: Cesarean Delivery; Uterine Contractility
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methyl-Ergonovine-Oxytocin
Drug: Oxytocin

SUMMARY:
Despite of marked improvements in clinical management, early postpartum hemorrhage(PPH)remains a significant contributor to maternal morbidity and mortality both in developing countries and in hospitals equipped with all that modern medicine has to offer. This complication is amongst the most challenging that a clinician will face in the obstetric patient. Prevention, early recognition and prompt appropriate intervention are the keys to minimizing the impact of PPH on women's health.

Patients undergoing Cesarean sections following failure to progress in labor are at great risk for PPH and should theoretically benefit from an additional uterotonic agent. This study will be conducted to define whether the addition of ergonovine maleate to oxytocin, administered in a prophylactic way, reduces blood loss during Cesarean section for failure to progress in labor.

DETAILED DESCRIPTION:
Despite of marked improvements in management, early postpartum hemorrhage(PPH)remains a significant contributor to maternal morbidity and mortality both in developing countries and in hospitals equipped with all that modern medicine has to offer. This complication is amongst the most challenging that a clinician will face in Obstetrics. Prevention, early recognition and prompt appropriate intervention are the keys to minimizing the impact of PPH on women's health.

Prophylactic oxytocin, commonly administered after fetal and placental delivery, has been shown to reduce the incidence of PPH. The main advantages of this drug are its rapid onset of action and the fact that it does not cause elevations of blood pressure or tetanic contractions like ergonovine. The effect of oxytocin is limited by the number and status of the oxytocin receptors. Increases in the dose of oxytocin will not necessarily improve uterine contraction, if receptors are not adequate in quantity and quality.This is the cause of patients exposed to oxytocin for labor augmentation, in whom oxytocin receptors are known to reduce both number and response to oxytocin. Therefore, a different uterotonic agent, involving a different mechanism of action should be used instead. Alternative drugs include ergot derivatives and prostaglandins (carboprost and misoprostol). Although protection from PPH with ergot derivatives and prostaglandin appear to be similar, prostaglandins are associated with more side effects.

Patients undergoing Cesarean sections following failure to progress in labor are at great risk for PPH and should theoretically benefit from an additional uterotonic agent. This study will be conducted to define whether the addition of ergonovine maleate to oxytocin, administered in a prophylactic way, reduces blood loss during Cesarean section for failure to progress in labor.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section secondary to failure to progress in labour
* First stage of labour
* Received oxytocin for at least 4 hours

Exclusion Criteria:

* Require General Anesthesia
* Cardiac Disease
* Hypertension
* Predisposition to uterine atony and postpartum hemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Blood loss | During surgery

SECONDARY OUTCOMES:
Effectiveness of Uterine Contraction | During surgery
Side Effects | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Balki M, Dhumne S, Kasodekar S, Kingdom J, Windrim R, Carvalho JC. Oxytocin-ergometrine co-administration does not reduce blood loss at caesarean delivery for labour arrest. BJOG. 2008 Apr;115(5):579-84. doi: 10.1111/j.1471-0528.2007.01658.x. PMID 18333937